CLINICAL TRIAL: NCT00280150
Title: Phase I/II Trial of Induction Carboplatin/Paclitaxel With Bevacizumab Followed by Concurrent Thoracic Conformal Radiation Therapy With Carboplatin/Paclitaxel, Bevacizumab and Erlotinib in Stage IIIA/B Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy, Bev, RT, and Erlotinib in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0511; UNC IRB 05-2091
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Erlotinib Hydrochloride; Paclitaxel; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Bevacizumab 10 mg + Chemoradiotherapy (carboplatin, paclitaxel, and 3-dimensional conformal radiation therapy)
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: paclitaxel; Radiation: 3-dimensional conformal radiation therapy
- Cohort 2 (Experimental): Bevacizumab 10 mg + Erlotinib 100 mg + Chemoradiotherapy (carboplatin, paclitaxel, and 3-dimensional conformal radiation therapy)
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: erlotinib hydrochloride; Drug: paclitaxel; Radiation: 3-dimensional conformal radiation therapy
- Cohort 3 (Experimental): Bevacizumab + Erlotinib 150 mg + Chemoradiotherapy (carboplatin, paclitaxel, and 3-dimensional conformal radiation therapy)
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: erlotinib hydrochloride; Drug: paclitaxel; Radiation: 3-dimensional conformal radiation therapy
- Phase II (Experimental): Bevacizumab + Erlotinib 100 mg + Chemoradiotherapy (carboplatin, paclitaxel, and 3-dimensional conformal radiation therapy)
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: erlotinib hydrochloride; Drug: paclitaxel; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Biological: bevacizumab — Given IV
Drug: carboplatin — Given IV
Drug: erlotinib hydrochloride — Given orally
  Arms: Cohort 2; Cohort 3; Phase II
Drug: paclitaxel — Given IV
Radiation: 3-dimensional conformal radiation therapy — Given 5 days a week for 7 weeks

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Radiation therapy uses high energy x-rays to kill tumor cells. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy together with bevacizumab, radiation therapy, and erlotinib may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of bevacizumab and erlotinib when given together with combination chemotherapy and radiation therapy and to see how well they work in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of bevacizumab and erlotinib hydrochloride when given together with carboplatin, paclitaxel, and thoracic conformal radiotherapy in patients with stage IIIA or IIIB non-small cell lung cancer. (Phase I [closed to accrual as of 1/3/2008])
* Determine the safety and toxicity profile of this regimen in these patients. (Phase I [closed to accrual as of 1/3/2008])
* Determine the progression-free survival of patients treated with induction therapy comprising carboplatin, paclitaxel, and bevacizumab followed by chemoradiotherapy comprising thoracic conformal radiotherapy, carboplatin, paclitaxel, bevacizumab, and erlotinib hydrochloride and consolidation therapy comprising bevacizumab and erlotinib hydrochloride. (Phase II)
* Determine the overall toxicity profile of this regimen in these patients. (Phase II)

Secondary

* Determine the response rate in patients treated with induction therapy comprising carboplatin, paclitaxel, and bevacizumab. (Phase I[closed to accrual as of 1/3/2008] and II)
* Determine the toxicity profile of induction therapy in these patients. (Phase I [closed to accrual as of 1/3/2008] and II)
* Determine the overall response rate and survival profile in patients treated with this regimen. (Phase I [closed to accrual as of 1/3/2008] and II)
* Determine the feasibility and tolerability of administering consolidation therapy comprising erlotinib hydrochloride and bevacizumab after treatment with combined modality therapy (induction therapy and chemoradiotherapy) in these patients. (Phase I [closed to accrual as of 1/3/2008] and II)
* Collect tumor and blood samples from these patients for future analysis of correlation between molecular markers and clinical benefit. (Phase I [closed to accrual as of 1/3/2008] and II)

OUTLINE: This is a nonrandomized, open-label, controlled, phase I (closed to accrual as of 1/3/2008), dose-escalation study of bevacizumab and erlotinib hydrochloride, followed by a phase II study.

* Phase I (closed to accrual as of 1/3/2008):

  * Induction therapy: Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 2 courses. Patients with stable or responding disease proceed to chemoradiotherapy.
  * Chemoradiotherapy: Patients receive chemoradiotherapy according to their assigned dose cohort:

    * Cohort 1: Patients undergo thoracic conformal radiotherapy (TCRT) on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47. Patients also receive carboplatin IV and paclitaxel IV on days 1, 8, 15, 22, 29, 36, and 43 and bevacizumab IV over 30-90 minutes on days 1, 15, 29, and 43.
    * Cohort 2: Patients undergo TCRT and receive carboplatin, paclitaxel, and bevacizumab as in cohort 1. Patients also receive oral erlotinib hydrochloride on days 2-5, 9-12, 16-19, 23-26, 30-33, 37-40, and 44-47.
    * Cohort 3: Patients undergo TCRT and receive carboplatin, paclitaxel, and bevacizumab as in cohort 1. Patients also receive higher doses of oral erlotinib hydrochloride on days 2-5, 9-12, 16-19, 23-26, 30-33, 37-40, and 44-47.

Cohorts of 5 patients receive chemoradiotherapy as described above until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 (with grade 4 toxicity) or 3 (with grade 3 toxicity) of 5 patients experience dose-limiting toxicity.

Three to 6 weeks after completion of chemoradiotherapy, patients proceed to consolidation therapy.

* Consolidation therapy: Patients receive bevacizumab IV on day 1 and oral erlotinib hydrochloride on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

  * Phase II:
* Induction therapy: Patients receive induction therapy as in phase I (closed to accrual as of 1/3/2008).
* Chemoradiotherapy: Patients undergo TCRT and receive carboplatin and paclitaxel as in phase I (closed to accrual as of 1/3/2008). Patients also receive bevacizumab and erlotinib hydrochloride as in phase I (closed to accrual as of 1/3/2008) at the MTD/drug combination determined in phase I (closed to accrual as of 1/3/2008).
* Consolidation therapy: Patients receive consolidation therapy as in phase I (closed to accrual as of 1/3/2008).

Tumor tissue and peripheral blood is collected at baseline for future correlative and biomarker studies.

After completion of study therapy, patients are followed every 2 months for 2 years, every 4 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer

  * Stage IIIA or IIIB disease
  * No malignant pleural or pericardial effusions
  * No palpable supraclavicular adenopathy
* Squamous cell histology allowed provided there is no hemoptysis and no central invasive lesions that abut or invade major blood vessels in the chest (with or without cavitation)
* Considered suitable and appropriate for combined modality therapy and thoracic conformal radiotherapy, as determined by the treating medical and radiation oncologist

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Hemoglobin ≥ 9.0 mg/dL
* Platelet count ≥ 100,000/mm³
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Forced expiratory volume 1 (FEV_1) ≥ 1 L
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≤ 2.5 times ULN
* Bilirubin normal
* Partial thromboplastin time (PTT) and international normalized ratio (INR) normal
* Urine protein:creatinine ratio < 1.0
* Blood pressure ≤ 150/100 mm Hg on 3 separate occasions
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant recent hemoptysis (> ½ teaspoon of bright red blood)
* No unstable angina
* No New York Heart Association (NYHA) congestive heart failure ≥ class II
* No myocardial infarction or stroke within the past 6 months
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious, non-healing wound, ulcer, or bone fracture
* No thrombosis requiring therapeutic anticoagulation
* No significant traumatic injury within the last 28 days

PRIOR CONCURRENT THERAPY:

* Recovered from prior surgery
* At least 4 weeks since prior and no concurrent participation in another experimental drug study
* At least 4 weeks since prior and no concurrent major surgical procedure or open biopsy
* At least 2 weeks since prior mediastinoscopy or mediastinotomy
* At least 1 week since prior fine needle aspirations or core biopsies
* No other concurrent antineoplastic or antitumor agents, including chemotherapy, radiotherapy, immunotherapy, or hormonal anticancer therapy
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-01; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Stinchcombe, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Thomas A. Stinchcombe, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina

REFERENCES:
- [Result] Socinski MA, Stinchcombe TE, Moore DT, Gettinger SN, Decker RH, Petty WJ, Blackstock AW, Schwartz G, Lankford S, Khandani A, Morris DE. Incorporating bevacizumab and erlotinib in the combined-modality treatment of stage III non-small-cell lung cancer: results of a phase I/II trial. J Clin Oncol. 2012 Nov 10;30(32):3953-9. doi: 10.1200/JCO.2012.41.9820. Epub 2012 Oct 8. PMID 23045594
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from four institutions between February 2006 and April 2010.
Pre-assignment Details: Of the 48 participants screened for eligibility, 46 were deemed eligible and went on to treatment, 1 was ineligible, and 1 was initially ruled eligible but the liver functioning tests (LFTs) continued to increase so the PI felt the participant should not be treated.
Groups:
- Cohort 1: Bevacizumab 10 mg + Chemoradiotherapy
- Cohort 2: Bevacizumab 10 mg + Erlotinib 100 mg + Chemoradiotherapy
- Cohort 3: Bevacizumab 10 mg + Erlotinib 150 mg + Chemoradiotherapy
- Phase II: Bevacizumab + Erlotinib 100 mg + Chemoradiotherapy
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Started | 5 | 5 | 6 | 30
Cohort Induction | 5 | 5 | 6 | 30
Consolidation Therapy | 2 | 5 | 3 | 0 (Phase II participants did not receive consolidation therapy.)
Completed | 2 | 4 | 1 | 20
Not Completed | 3 | 1 | 5 | 10
Not completed — Adverse Event | 0 | 1 | 2 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Did not get consolidation therapy | 3 | 0 | 3 | 0
Not completed — Declining Performance Status | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase II: Bevacizumab + Erlotinib100 mg + Chemoradiotherapy (carboplatin, paclitaxel, and 3-dimensional conformal radiation therapy)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II | Total
Number analyzed (Participants) | 5 | 5 | 6 | 30 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 3 | 18 | 28
  >=65 years | 1 | 2 | 3 | 12 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 16 | 22
  Male | 4 | 3 | 3 | 14 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 5 | 6 | 29 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 7 | 10
  White | 4 | 4 | 4 | 22 | 34
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 6 | 30 | 46

OUTCOME MEASURES:

1. Primary Outcome: Maximum Dose of Erlotinib When Given Together With Carboplatin, Paclitaxel, and Thoracic Conformal Radiotherapy (Phase I [Closed to Accrual as of 1/3/2008])
Description: Dose-limiting toxicities (DLTs) were used to establish which cohort would be used for the phase II portion of the trial. DLTs were defined as any grade 3 or 4 nonhematologic toxicity with the exception of esophagitis, which had to be grade 4; grade 4 neutropenia lasting greater than or equal to 7 days and thrombocytopenia to less than 20,000/microliter.
Time Frame: 6 weeks after completion of therapy
Population: This was a phase I objective only, so the phase II participants are not included.
Measure: Number; unit: DLTs
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 5 | 5 | 6 | 0
DLTs | 0 | 0 | 2 |

2. Primary Outcome: Safety and Toxicity Profile of Combining Both Bevacizumab and Erlotinib Hydrochloride With Carboplatin, Paclitaxel, and Thoracic Conformal Radiotherapy
Description: A list of Hematologic and nonhematologic toxicities associated with induction and concurrent therapy. This includes the percentage of patients who experienced grades 2-4 based on the National Cancer Institute Common Terminology Criteria for Adverse Events (version 3.0).
Time Frame: 6 weeks after completion of therapy
Population: Of the 46 patients, one was retrospectively diagnosed as having stage IV NSCLC after induction therapy was withdrawn from the protocol therapy leaving 45 evaluable for toxicity. 42 patients were eligible for concurrent therapy.
Measure: Number; unit: percentage of participants
Groups:
- Induction Therapy: Percentage of all patients receiving induction therapy
- Concurrent Therapy: Percentage of all patients receiving concurrent therapy
Arm/Group | Induction Therapy | Concurrent Therapy
Number analyzed (Participants) | 45 | 42
percentage of participants
  Anemia | 4 | 17
  Neutrophenia | 52 | 35
  Thrombocytopenia | 0 | 16
  Febrile neutropenia | 0 | 2
  Nausea/vomiting | 7 | 6
  Fatigue | 20 | 22
  Alopecia | 42 | 9
  Hypertension | 9 | 4
  Myalgias/arthralgias | 27 | 0
  Diarrhea | 6 | 2
  Neuropathy | 2 | 2
  Rash | 2 | 11
  Anorexia | 0 | 6
  Esophagitis | 0 | 40
  Dehydration | 0 | 11
  Hemorrhage | 0 | 6
  Hypomagnesemia | 0 | 4
  Proteinuria | 0 | 2
  Weight loss | 0 | 9
  Pneumonitis | 0 | 2
  Hypersensitivity reaction | 4 | 2

3. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time during and after the treatment of a stage IIIA/B NSCLC that a patient lives with the disease but it does not get worse. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 5 years
Population: Of the 46 patients, one was retrospectively diagnosed as having stage IV NSCLC after induction therapy was withdrawn from the protocol therapy leaving 45 evaluable patients.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Overall Study: This includes patients from all cohorts.
Arm/Group | Overall Study
Number analyzed (Participants) | 45
Months | 10.2 [8.4 to 18.3]

4. Secondary Outcome: Response Rate to Induction Therapy (Phase I [Closed to Accrual as of 1/3/2008] and II)
Description: Measurable lesions must be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10mm with spiral CT scan or nonmeasurable, but evaluable. Evaluable is nonmeasurable disease that includes ascites, malignant pleural/pericardial effusion, bone lesions, or marrow involvement. The same method of assessment and the same techniques should be used to characterize each identified and reported lesion at baseline and during follow-up.
  Complete Response (CR)- Disappearance of all target lesions
Time Frame: 5 years
Population: 43 of 45 patients received both cycles of induction C/P therapy plus bevacizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 43
Participants | 0

5. Secondary Outcome: Overall Response Rate and Survival Profile
Description: The overall response rate (ORR) to the two cycles of induction therapy plus bevacizumab in stage IIIA/B NSCLC. ORR is the portion of patients with a tumor size reduction for a minimum time period. Response duration is measured from the time of initial response until documented tumor progression.
Time Frame: 5 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Overall Study: All 45 patients were included in the summary of efficacy outcomes.
Arm/Group | Overall Study
Number analyzed (Participants) | 45
percentage of participants | 39 [24 to 55]

6. Secondary Outcome: Feasibility and Tolerability of Administering Consolidation Therapy
Description: The proportion of patients who were able to complete consolidation therapy after induction therapy and chemoradiotherapy
Time Frame: 6 cycles
Population: Of the initial 14 patients, only 9 (64%) patients were able to start consolidation therapy and only 5 (36%) patients were able to complete 6 cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 14
Participants | 5

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Overall Study: Of the 46 patients, one was retrospectively diagnosed as having stage IV NSCLC after induction therapy was withdrawn from the protocol therapy leaving 45 evaluable patients. This includes patients from all cohorts.
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 30/45
Serious Adverse Events (participants affected / at risk) | 19/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=45)
Esophagitis (Gastrointestinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Bronchus (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage/Bleeding - Other (Specify, __) (Vascular disorders) | 1
Pain - Chest/thorax NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Esophagitis (Gastrointestinal disorders) | 5
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 2
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1
Infection with unknown ANC - Esophagus (Infections and infestations) | 2
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1
Neurology - Other (Specify, __) (Nervous system disorders) | 1 — Neurotoxicity-sensory neuropathy
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Rigors/chills (General disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=45)
Alkaline phosphatase (Investigations) | 2
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 6
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 12
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 3
Burn (Injury, poisoning and procedural complications) | 1
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Creatinine (Investigations) | 4
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Diarrhea (Gastrointestinal disorders) | 18
Dizziness (Nervous system disorders) | 8
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 7
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6
Edema: head and neck (General disorders) | 1
Edema: limb (General disorders) | 2
Esophagitis (Gastrointestinal disorders) | 27
Extremity-lower (gait/walking) (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 34
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Flushing (Vascular disorders) | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 1 — Odynophagia
Glomerular filtration rate (Renal and urinary disorders) | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 35
Heartburn/dyspepsia (Gastrointestinal disorders) | 6
Hematoma (Vascular disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 22
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 5
Hemorrhage, GU - Bladder (Renal and urinary disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 13
Hemorrhage/Bleeding - Other (Specify, __) (Vascular disorders) | 6
Hemorrhoids (Gastrointestinal disorders) | 1
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes/flushes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 10
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 3
Infection - Other (Specify, __) (Infections and infestations) | 2
Infection (Infections and infestations) | 2 — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Esophagus
Infection with normal ANC or Grade 1 or 2 neutrophils - Foreign body (Infections and infestations) | 1 — e.g., graft, implant, prosthesis, stent
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1
Infection with unknown ANC - Esophagus (Infections and infestations) | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1
Infection with unknown ANC - Sinus (Infections and infestations) | 2
Injection site reaction/extravasation changes (General disorders) | 1
Insomnia (Psychiatric disorders) | 4
Joint-function (Metabolism and nutrition disorders) | 1
Leukocytes (total WBC) (Investigations) | 7
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 7
Metabolic/Laboratory - Other (Specify, __) (Investigations) | 3
Mood alteration - Anxiety (Psychiatric disorders) | 1
Mood alteration - Depression (Psychiatric disorders) | 1
Mucositis/stomatitis (clinical exam) - Esophagus (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5
Mucositis/stomatitis (functional/symptomatic) - Esophagus (Gastrointestinal disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Extraocular (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 18
Neurology - Other (Specify, __) (Nervous system disorders) | 2
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 21
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 34
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 6
Pain - Bone (Musculoskeletal and connective tissue disorders) | 2
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain - Chest/thorax NOS (General disorders) | 2
Pain - Esophagus (Gastrointestinal disorders) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 24
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 15
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1
Pain - Oral-gums (Gastrointestinal disorders) | 2
Pain - Other (Specify, __) (General disorders) | 2
Pain - Pain NOS (General disorders) | 2
Pain - Rectum (Gastrointestinal disorders) | 1
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 3
Platelets (Investigations) | 20
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Proteinuria (Renal and urinary disorders) | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 12
Rash: dermatitis associated with radiation - Chemoradiation (Injury, poisoning and procedural complications) | 4
Rash: dermatitis associated with radiation - Radiation (Injury, poisoning and procedural complications) | 3
Renal failure (Renal and urinary disorders) | 1
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 1 — Urinary burning
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Stricture/stenosis (including anastomotic), GI - Esophagus (Gastrointestinal disorders) | 9
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 5
Ulcer, GI - Esophagus (Gastrointestinal disorders) | 7
Ulceration (Skin and subcutaneous tissue disorders) | 1
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 1
Vision-blurred vision (Eye disorders) | 2
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 9
Weight loss (Investigations) | 7
Mental Status (Nervous system disorders) | 1
Gastrointestinal - Other (Specify,___) (Gastrointestinal disorders) | 1 — Oral Abcess

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days